CLINICAL TRIAL: NCT00984568
Title: Conventional Step-Up Versus Infliximab Monotherapy in Patients With Active Moderate to Severe Ulcerative Colitis. A Randomized, Open Label, Prospective, Multicenter Study
Brief Title: Conventional Step-Up Versus Infliximab Monotherapy in Patients With Ulcerative Colitis (P05553)
Acronym: MUNIX
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to slow recruitment the study was stopped prematurely.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05553; 2009-010065-23 (EudraCT Number)
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Results first posted 2013-04-02 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Infliximab; Prednisolone; Prednisone; Mesalamine; Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Top-Hold (Experimental): Level 1: Infliximab IV 5 mg/kg at Weeks 0, 2, and 6, and every 8 weeks thereafter. Level 2: Infliximab IV 5 mg/kg every 4 weeks. Level 3: Prednisolone induction + AZA 2.0-2.5 mg/kg/day.
  Interventions: Biological: Infliximab; Drug: Prednisolone; Drug: Azathioprine
- Step-Up (Active Comparator): Level 1: Oral prednisolone (40 mg/day or 1 mg/kg/day in the case of non-response) + oral 5-aminosalicylic acid (5-ASA) 2 g/day. Level 2: Oral prednisolone (40 mg/day or 1 mg/kg/day in the case of non-response) + oral azathioprine (AZA) at a dose of 2.0-2.5 mg/kg/day. Level 3: Infliximab 5 mg/kg at Weeks 0, 2, and 6 and every 8 weeks thereafter.
  Interventions: Biological: Infliximab; Drug: Prednisolone; Drug: 5-aminosalicylic acid; Drug: Azathioprine

INTERVENTIONS:
Biological: Infliximab — Infliximab intravenous infusion at a dose of 5 mg/kg.
  Other Names: Remicade; SCH 215596
Drug: Prednisolone — Oral prednisolone 40 mg/day or 1 mg/kg/day depending upon participant response.
  Other Names: Decortin
Drug: 5-aminosalicylic acid — 5-ASA administered orally at a dose of 2 g/day.
  Other Names: 5-ASA; Pentasa
  Arms: Step-Up
Drug: Azathioprine — AZA administered orally at a dose of 2.0-2.5 mg/kg/day.
  Other Names: AZA; Imurek

SUMMARY:
This study will be performed to compare the efficacy and safety of the classical "Step-Up" approach for treatment of moderate-to-severe active ulcerative colitis using oral prednisolone + oral 5-aminosalicylic acid (5-ASA) or oral prednisolone + oral azathioprine (AZA) with a more intensive and early "Top-Hold" approach with intravenous infliximab (5 mg/kg) administered at Weeks 0, 2, and 6 and 8 weeks thereafter.

DETAILED DESCRIPTION:
Participants will be randomized to receive either intravenous (IV) infliximab monotherapy (Top-Hold approach) starting at a dose of 5 mg/kg at Weeks 0, 2, and 6 and thereafter every 8 weeks in Level 1, or classical Step-Up treatment starting with oral prednisolone (40 mg/day for at least 3 days and at most 2 weeks followed by 1 mg/kg/day for a minimum of 7 days and up to 2 weeks in the case the participant does not show an improvement in clinical symptoms under 40 mg/day treatment) + oral 5-aminosalicylic acid (5-ASA) at a dose of 2 g/day in Level 1.

Participants receiving Step-Up treatment who have not achieved adequate response during the first 4 weeks of prednisolone treatment will directly enter Level 3 treatment after endoscopy is performed to confirm treatment eligibility. Furthermore, participants that have not achieved response at Week 4 will also directly enter Level 3 and be switched to treatment with IV infliximab.

If a participant experiences a first flare after initial response, participants in the Step-Up group will start prednisolone treatment at the last effective dose (i.e., participants that previously responded to prednisolone 40 mg/day will receive a dose of 40 mg/day for at least 3 days and up to 2 weeks; participants that previously responded to prednisolone 1 mg/kg/day will receive a dose of 1 mg/kg/day for a minimum of 7 days and up to 2 weeks). If the last effective dose was 40 mg/day and the participant does not respond within 14 days, the dose will be adjusted to 1 mg/kg/day for a minimum of 7 days and up to 2 weeks. In case the participant does not respond to prednisolone (i.e., does not return to their individual baseline partial Mayo score obtained at study Week 4), the participant will enter Level 3 and receive treatment with IV infliximab.

If a participant experiences a second flare after initial response at Week 4 (Level 1), the participant will enter treatment Level 2. In Level 2, participants will receive a prednisolone induction at the same effective dose as previously used in Level 1 + maintenance treatment with oral azathioprine (AZA) at a dose of 2.0-2.5 mg/kg/day. Participants that do not respond to this treatment at Level 2 or that develop a further flare after initial response at Level 2 will enter Level 3 and will receive treatment with IV infliximab following endoscopy to confirm treatment eligibility.

If at any time during treatment, a participant becomes prednisolone dependent (i.e., flare during tapering phase of prednisolone), the participant will enter Level 3 treatment with IV infliximab.

Participants in Level 1 of the Top-Hold treatment group (IV infliximab at Week 0, 2, and 6 and every 8 weeks thereafter) that have not achieved response at Week 4 will receive IV infliximab 5 mg/kg at reduced intervals of 4 weeks (Level 2) starting with the Week 10 infusion. Participants suffering a flare after initial response in Level 1 will be switched to to Level 2. Participants that do not respond to treatment at reduced intervals after 3 infusions (12 weeks), or that develop a further flare after initial response at Level 2, will be switched to treatment with oral prednisolone + AZA (Level 3) following colonoscopy to confirm eligibility.

When a participant responds to treatment with IV infliximab in Level 2, they will return to treatment with IV infliximab every 8 weeks when response is achieved at 3 consecutive visits.

ELIGIBILITY:
Inclusion Criteria:

* Any race or ethnicity
* Must have a diagnosis of moderate-to-severe active ulcerative colitis (UC) with inflammation present beyond the rectum and including more than 20 cm of the colon (Mayo score of 6 to 12 points, inclusive ≥ 2 in the endoscopy subscore)
* Must have responded inadequately to oral (with or without topical) 5-ASA treatment (prerequisite oral: at a minimum 4 g/d for 7 days) and must be considered for the first course of systemic corticosteroids; Participants with a UC and a Mayo score of ≥ 9 are also eligible without prior 5-ASA treatment
* Must agree to use acceptable methods of contraception for at least 2 weeks prior to starting any study treatment and to continue until at least 6 months after the last doses of study drugs
* Laboratory results must be within specified limits
* Must be negative for colorectal cancer or any associated lesions
* Must have a negative tuberculosis (TB) test
* Must have a chest x-ray within the 3 months with no clinically significant abnormality, or evidence of current active TB or latent TB
* Must have a negative stool culture

Exclusion Criteria:

* Pregnant, nursing, or planning pregnancy
* Had received previous treatment for UC with the corticosteroids, infliximab, azathioprine/

  6-mercaptopurine (6-MP), cyclosporine, tacrolimus, methotrexate, sirolimus, mycophenolate, any tumor necrosis factor-alpha (TNF-α) inhibitor or receptor constructs that bind to ΤΝF-α (e.g., etanercept or adalimumab) and any other biologic agents
* Frequent (chronic) use of non-steroidal anti-inflammatory drugs (NSAIDs)
* Use of laxatives or any murine recombinant product
* Had surgery for active gastrointestinal bleeding, peritonitis, intestinal obstruction, or intra-abdominal or pancreatic abscess requiring surgical drainage in previous 2 months
* History of colonic obstruction within the previous 6 months
* History of mucosal dysplasia, fistula or colonic resection, adenomatous polyps or stoma, severe, fixed symptomatic stenosis of the large or small intestine
* Had serious infection with previous 2 months, including human immunodeficiency virus (HIV) and hepatitis
* Had organ transplant (with the exception of a corneal transplant)
* Any malignancy within 5 years, including lymphoma
* History of demyelinating disease such as multiple sclerosis or optic neuritis
* Presence or history of congestive heart failure
* Requires chronic and frequent use of antimotility agents for control of diarrhea
* Requires total parenteral nutrition
* Had participated in any other clinical trial within 30 days or intention to participate in another clinical trial during participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Hasskamp J, Meinhardt C, Patton PH, Timmer A. Azathioprine and 6-mercaptopurine for maintenance of remission in ulcerative colitis. Cochrane Database Syst Rev. 2025 Feb 27;2(2):CD000478. doi: 10.1002/14651858.CD000478.pub5. PMID 40013523

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Top-Hold | Step-Up
Started | 15 | 13
Completed | 7 | 7
Not Completed | 8 | 6
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lack of Efficacy | 2 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Did Not Meet Randomization Criteria | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Opportunistic Infection | 1 | 0
Not completed — Unknown Reason | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Top-Hold | Step-Up | Total
Number analyzed (Participants) | 15 | 13 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (15.2) | 41.6 (15.3) | 40.7 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 5 | 6 | 11

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants Achieving Treatment Response
Description: Response was defined as a minimum decrease from baseline in total Mayo score of 3 points and 30% up to and including 4 weeks after the start of treatment. The Mayo score consists of the following 4 subscores: stool frequency; rectal bleeding; endoscopy results; physician's global assessment. Each subscore
  is rated on a scale from 0 (best) to 3 (worst). The total Mayo score is calculated as the sum of the 4 subscores and ranges from 0 (best) to 12 (worst).
Time Frame: Up to Week 4
Population: The full analysis set (FAS) consisted of all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Top-Hold | Step-Up
Number analyzed (Participants) | 15 | 13
Participants | 10 | 10

2. Primary Outcome: Number of Participants With Response at Week 4 and Steroid-Free Remission at Week 50
Description: Response at Week 4 was defined as a minimum decrease from baseline in Mayo score of 3 points and 30%. Steroid-free remission at Week 50 was defined as a total Mayo score (including endoscopic assessment) of 2 points or lower and no individual subscore exceeding 1. The Mayo score consists of the following 4 subscores: stool frequency; rectal bleeding; endoscopy results; physician's global assessment. Each subscore is rated on a scale from 0 (best) to 3 (worst). The total Mayo score is calculated as the sum of the 4 subscores and ranges from 0 (best) to 12 (worst).
Time Frame: Week 50
Population: The FAS consisted of all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Top-Hold | Step-Up
Number analyzed (Participants) | 15 | 13
Participants | 5 | 5

ADVERSE EVENTS:
Time Frame: Up to Week 50
Arm/Group | Top-Hold | Step-Up
Serious Adverse Events (participants affected / at risk) | 2/15 | 1/13
Other Adverse Events (participants affected / at risk) | 14/15 | 11/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Top-Hold (N=15) | Step-Up (N=13)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Top-Hold (N=15) | Step-Up (N=13)
Nasopharyngitis (Infections and infestations) | 4 (4) | 6 (6)
Gastrointestinal Viral Infection (Infections and infestations) | 0 (0) | 2 (2)
Borrelia Infection (Infections and infestations) | 1 (1) | 0 (0)
Candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Clostridial Infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis Astroviral (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis Norovirus (Infections and infestations) | 1 (1) | 0 (0)
Giardiasis (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter Gastritis (Infections and infestations) | 0 (0) | 1 (1)
Herpes Simplex (Infections and infestations) | 0 (0) | 1 (1)
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (2)
Scarlet Fever (Infections and infestations) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (4)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis Ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis Erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Periodontitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Reflux Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muskuloskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (3) | 1 (1)
Infusion Related Reaction (General disorders) | 1 (9) | 1 (2)
Oedema Peripheral (General disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (3)
Intercostal Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Sensory Loss (Nervous system disorders) | 1 (1) | 0 (0)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cushing's Syndrome (Endocrine disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Coombs Test Positive (Investigations) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Aortic Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to slow recruitment the study was stopped prematurely; participants on study at that time continued to receive treatment per protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide the sponsor 45 days prior to publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial. The sponsor has the right to review and comment with respect to publications, abstracts, slides, and manuscripts and the right to review and comment on the data analysis with respect to: proprietary information, accuracy, and fair balance.